CLINICAL TRIAL: NCT04504968
Title: Randomized Clinical Trial to Evaluate the Effectiveness of a Multimodal Intervention Program in Prefrail and Frail Type 2 Diabetic Patients on Frailty and Quality of Life in Latinamerican Countries
Brief Title: Effectiveness of a Multimodal Intervention on Function in Older Frail People With Diabetes in Latinamerican
Acronym: DIABFRAIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Collaborators: Pan American Health Organization (Other); Catholic University of the Sacred Heart (Other); Diabetes Frail Ltd (Other); University of Castilla-La Mancha (Other); Confederación Española de Organizaciones de Mayores (CEOMA) (Unknown); Pontificia Universidad Javeriana (Other); Pontificia Universidad Catolica de Chile (Other); Instituto Nacional de Geriatria, Mexico (Other Government); Universidad de San Martín de Porres (USMP) (Unknown); Universidad de Santiago de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIABFRAIL-LATAM
Record Dates: First submitted 2020-05-05; First posted 2020-08-07 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Frailty Syndrome; Frail Elderly Syndrome; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Frailty; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: he DIABFRAIL-LATAM is an open randomized clinical trial, with random allocation 1:1 by participants to Usual Care Group (UCG) or Intervention Group (IG)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Multimodal intervention:
  Interventions: Other: Multimodal intervention
- Usual care group (Placebo Comparator): Usual care group
  Interventions: Other: Usual care group

INTERVENTIONS:
Other: Multimodal intervention — 1. Optimal control: HbA1c between 7.6-8.5% (60-69 mmol/mol) and Blood Pressure<150/90 mmHg
  2. The physical exercise program that will be used will be the Vivifrail program (Erasmus + UE). Vivifrail includes: Strength for arms and legs, balance and gait, flexibility and resistance. The duration will be 16 weeks. (3 weeks to explain the program in the Trial site and the rest of weeks, it will be carried out at home).
  3. Nutritional and educational program to increase diabetes knowledge, develop practical self-care skills for diabetes and increase the likelihood of improving glycemic control safely. The intervention aims to minimize the risk of hypoglycemia, ensure optimal nutritional status and help to maintain functional status. Seven separate sessions of 45 minutes each one twice a week for a period of 3-4 weeks in small groups. They will be moderated by a physician or diabetes educator and focused on behavioral changes and key points.
  Arms: Intervention group
Other: Usual care group — The level of usual health care that a patient with diabetes receives from their local national health system
  Arms: Usual care group

SUMMARY:
Randomized clinical trial, international, multicentre, single-blind, two parallel groups, pragmatic. It will be carried out by investigators in several Latin American countries (Chile, Colombia, Mexico and Peru) and with random allocation 1:1 of the participants to Usual Care Group (UCG) or Intervention Group (IG). Each country will select 5 trial sites that will recruit 0-60 participants. Finally, 1050 subjects will be involved in the project.

The primary outcome are the changes in function and quality of life as measured by changes in the scores used to assess them between baseline and 1-year follow-up. Function will be assessed by the Short Physical Performance Battery-SPPB.

This study is focused on an older population (≥ 65 years) with diabetes and a frail or prefrail status

The intervention includes:

Educational program in small groups: 7 sessions in the clinical trial sites (2 sessions a week for the first 3-4 weeks) Exercise program (16 weeks): learning phases in clinical trial site for 3-4 first week (coincident with the educational program sessions) and the rest at home.

Adaptation of targets of HbA1c and blood pressure (BP). UCG Usual care group consists in level of care usually given in Health Care system.

DETAILED DESCRIPTION:
International, multicentre, single-blind, two parallel groups, pragmatic randomised Research Clinical Trial. It will be carried out by investigators in several Latin American countries (Chile, Colombia, Mexico and Peru) and with random allocation 1:1 of the participants to Usual Care Group (UCG) or Intervention Group (IG). Each country will select 5-7 trial sites that will recruit 51 participants (255 participants per country) except Mexico which will select 2 sites to recruit 50 participants each one (100 participants).

There will be a National lead investigator in each involved country. This National lead investigator will be trained by the general coordinator team in the procedures of the study. Each National lead investigator will be responsible for the training in his/her country. In each country, the lead will select the recruitment trial sites (5-7 in each country) and each trial site will recruit 51 participants approximately except in Mexico (see above). All data will be collected in an eCRF (electronic case report form) platform designed specifically for this project.

This study is focused on an older population (≥ 65 years) with diabetes and a frail or prefrail status.

Objectives:

Main objective: To assess the effectiveness of a multi-modal intervention in subjects with type 2 Diabetes Mellitus aged ≥ 65 years who are frail or pre-frail in terms of function and quality of life in comparison with usual clinical practice.

Secondary objectives:

* Changes in the frailty status (trajectories of frailty: frail to prefrail; frail to robustness; prefrail to robustness and vice versa).
* Incidence rate of symptomatic hypoglycemia and hypoglycemic coma.
* Incidence rate of hospital admission.
* Incidence rate of permanent institutionalization.
* Carer burden.
* Laboratory biomarkers of prognostic value for response to treatment

Usual care group:

Usual clinical practice is the level of usual health care that a patient with diabetes receives from their local national health system.

Intervention group:

1. Optimal glycosylated hemoglobin range between 7.6-8.5% (60-69 mmol/mol) and optimal blood pressure: <150/90 mmHg
2. Physical exercise program that will be used will be the Vivifrail program, developed in Europe (Erasmus + UE). Vivifrail includes:

   * Strength exercises for arms and legs.
   * Balance and gait, to avoid falls.
   * Flexibility.
   * Resistance. The duration of the training program will be 16 weeks.
3. Nutritional and educational program: The intervention is designed to increase diabetes knowledge, develop practical self-care skills for diabetes, and increase the likelihood of improving glycemic control safely. The intervention aims to minimize the risk of hypoglycemia, ensure optimal nutritional status, and help maintain functional status.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 65 years.
* The subject is willing and able to give written informed consent for participation in the study.
* Diagnosis of type 2 diabetes for at least 2 years
* Require to fulfill Fried´s criteria for frail or pre-frail individuals

Exclusion Criteria:

* Unable or unwilling to provide informed consent or accept randomization to either study group
* Plans to relocate out of the study area within the year or plans to be out of the study area for more than 6 consecutive weeks in the next year
* MoCA (Montreal Cognitive Assessment) lower than 17/30
* Cancer requiring treatment in the past 3 years,except for non-melanoma skin cancers or cancers that have an excellent prognosis (e.g., early stage breast or prostate cancer)
* Barthel ADL score lower than 60 points
* Inability to carry out the SPPB test (total score = 0)
* Upper and/or lower extremity amputation
* Current participation in a structured physical activity (PA) program, physical therapy or cardiopulmonary rehabilitation
* Current enrolment in another randomized clinical trial (RCT) involving lifestyle, nutrition, or pharmaceutical interventions
* Other medical, psychiatric, or behavioral factors that in the judgment of the investigator may interfere with the study participation
* Other illness of such severity that life expectancy is expected to be less than 12 months
* Any other condition that is an absolute contraindication to the exercise program:
* Acute heart attack (recent 3-6 months) or unstable angina
* Uncontrolled atrial or ventricular arrhythmias
* Aortic dissecting aneurysm
* Severe aortic stenosis
* Acute endocarditis / pericarditis
* Uncontrolled high blood pressure (> 180/100 mmHg)
* Acute thromboembolism
* Acute or severe heart failure
* Acute or severe respiratory failure
* Uncontrolled postural hypotension
* Uncontrolled acute decompensated diabetes mellitus or low blood sugar
* A recent fracture in the last month Any other circumstance the investigator believes to prevent undertaking physical activity

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 713 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Difference in physical function | 1 year
  (SPPB scale)The primary outcome is the difference in function after 12 months of follow-up between the intervention group and usual clinical practice measured by changes in the Short Physical Performance Battery (SPPB) scale. SPPB scores between 0-12. 0 is the worse and 12 the best value.

SECONDARY OUTCOMES:
Frailty trajectories | 1 year
  Trajectories of frailty according to changes in Fried´s phenotype. Frieds Phenotype scores between 0 and 5. 0 means robust; 1-2 mean prefrail and 3 or more mean frail
Frailty trajectories | 1 year
  Trajectories of frailty according to changes frail trait scale (FTS). FTS scores between 0-50. 0 is the best value and 50 the worst value.
Frailty trajectories | 1 year
  Trajectories of frailty according to changes in FRAIL scale. FRAIL scores SPPB scores between 0-5. 0 means robust; 1-2 mean prefrail and 3 or more mean frail
Basic activities of daily living | 1 year
  Deterioration of basic activities of daily living (BADL) according to changes in at least 10 points of Barthel index. Barthel scores between 0-100; 0 is the worst value and 100 the best.
Instrumental activities of daily living | 1 year
  Deterioration of instrumental activities of daily living (IADL) according to changes in at least 1 point of Lawton scale. Lawton scale scores between 0-10; 0 is the worst and 10 the best value
Rate of Hypoglycemia | 1 year
  Episodes of symptomatic hypoglycemia (proven glycaemia below 4mmol/L, or signs and symptoms attributed to hypoglycemia that respond to specific treatment) and hypoglycemic coma
Number of Hospital admission | 1 year
  Episodes of hospital admission (any overnight admission)
Number of patients with Permanent institutionalization | 1 year
  Permanent Institutionalization yeas or not
Rate of Falls | 1 year
  Number of falls
Rate of Severe Falls | 1 year
  Number of severe falls (2 or more falls in the year or at least 1 fall that requires medical assistance)
Caregiver burden | 1 year
  Caregiver burden (if exist) evaluated by the Zarit scale (ZBI). The ZBI consists of 22 items rated that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0-88.9 Higher scores indicate greater burden.
Rate of mortality | 1 year
  Number of patients who died
Health-related quality of life | 1 year
  Changes in Participant Health-related quality of life evaluated by EuroQoL 5D 3L(European Quality of life). EuroQoL scores between 0-10 and 10 is the worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: LEOCADIO RODRIGUEZ-MAÑAS, PhD, Principal Investigator — Consorcio Centro de Investigación Biomédica en Red (CIBER)
Locations (1):
- Hospital San Ignacio_Universidad Javeriana, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No